CLINICAL TRIAL: NCT02767518
Title: Does Prehabilitation Prior to Thoracic Aortic Repair Improve Quality of Care?
Brief Title: Prehabilitation for Aortic Repair Patients
Acronym: PREPARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Transfer of main study team to another institution
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dr. Bo Yang, Associate Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00109521
Record Dates: First submitted 2016-04-15; First posted 2016-05-10 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): Participants will be referred to the Michigan Surgical & Health Optimization Program in the month leading up to their surgery. Individuals are encouraged to increase their physical activity, practice stress reduction, and other behaviors associated with good health.
  Interventions: Behavioral: Prehabilitation
- Usual Care (No Intervention): Participants will follow the pre-operative instructions provided by their surgical team.

INTERVENTIONS:
Behavioral: Prehabilitation — Participants will receive an informational DVD, a pedometer, an incentive spirometer and access to the program website to help promote healthful behaviors and improved well-being in the days leading up to surgery.
  Other Names: MSHOP - Michigan Surgical & Health Optimization Program
  Arms: Prehabilitation

SUMMARY:
This is a 2-group study comparing the effect of a "prehabilitation" program to usual care on quality of life and clinical outcomes in patients undergoing elective repair of their thoracic aorta.

DETAILED DESCRIPTION:
Patients undergoing elective repair of their thoracic aortic aneurysm will be randomized to a "prehabilitation" program prior to their surgery or to usual care. The prehabilitation program is self-directed program designed to improve health and quality of life prior to surgery. The program is currently offered to general surgery patients; this study will examine the feasibility and acceptability of such a program in a different patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Diagnosis of thoracic aortic disease with scheduled repair
* Medical clearance from cardiothoracic surgeon
* Ability to provide informed consent
* Regular use of a smartphone or personal computer

Exclusion Criteria:

* Conditions that limit walking to a severe degree
* Current participation in regular physical activity program
* Acute aortic dissection
* Recent coronary artery disease events
* Inability to speak and read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting and enrolling | 1 year
  We will measure feasibility according to whether we are able to recruit and enroll subjects.

SECONDARY OUTCOMES:
Acceptability | 1 year
  We will ask patients to describe their experiences with the prehab program.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yang, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No